CLINICAL TRIAL: NCT03355612
Title: A Randomized, Multicenter, Controlled Study of XELOX (Oxaliplatin With Capecitabine) Combined With Apatinib Versus XELOX as Post-operative Chemotherapy in Locally Advanced Gastric Signet Ring Carcinoma With D2 Dissection.
Brief Title: XELOX Plus Apatinib vs XELOX as Post-operative Chemotherapy in Locally Advanced Gastric Signet Ring Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESAPAS Trial
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Gastric Carcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib; XELOX; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Drug:Apatinib with XELOX(Capecitabine and Oxaliplatin)
  Interventions: Drug: Apatinib; Drug: XELOX
- active comparator (Active Comparator): Drug:XELOX(Capecitabine and Oxaliplatin)
  Interventions: Drug: XELOX

INTERVENTIONS:
Drug: Apatinib — Apatinib: 500 mg, qd, po, last 180 days
  Other Names: YN968D1
  Arms: experimental group
Drug: XELOX — Capecitabine:1000 mg/m2 bid d1-14 q3w, Oxaliplatin:130 mg/m2 d1 q3w
  Other Names: Capecitabine and Oxaliplatin

SUMMARY:
This is a randomized, multicenter, controlled study to compared the Efficacy and Safety of XELOX combined with Apatinib versus XELOX as post-operative chemotherapy in locally advanced gastric signet ring carcinoma with D2 dissection.

DETAILED DESCRIPTION:
The purpose of this study is to prove that as for disease free survival time, and safety, Apatinib with XELOX(Oxaliplatin with Capecitabine) has a better effect over that of XELOX adjunct therapy group for postoperative chemotherapy of locally advanced gastric signet ring carcinoma with D2 dissection.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥ 18 and ≤ 70 years of age;
* 2. Eastern Cooperative Oncology Group Performance Status: 0-1;
* 3. Had been treated with Radical resection (D2, R0) of gastric cancer (Lymph node≥16);
* 4. Postoperative histological proven gastric signet-ring cell carcinoma(or contains signet-ring cell carcinoma);
* 5. Pathological stage:IIIA-IIIC（8th AJCC TNM）;
* 6. Patients have adequate baseline organ and marrow function :hemoglobin≥9g/dL; absolute neutrophil count (ANC) ≥1,500/mm3; PLT(platelets)≥1000,000/mm3; total bilirubin ≤1.5×upper normal limit(ULN); AST ≤2.5 ×ULN, ALT ≤2.5 ×ULN; prothrombin time-international normalized ratio≤1.5, and APTT(activated partial thromboplastin time) was within normal range; creatine ≤ 1.5 x ULN;
* 7. The ECG(electrocardiography) was basically normal in the 4 weeks before the study, and there was no obvious clinical symptoms of heart disease;
* 8. sign informed consent.

Exclusion Criteria:

* 1. Patients with hypertension and uncontrolled hypertension with hypotensive drugs therapy ;
* 2. Patients with dysphagia, complete or incomplete digestive tract obstruction, gastrointestinal bleeding, perforation, etc;
* 3. Patients had bradycardia or a QT extension;
* 4. Patients had gastrointestinal fistula and lacerations after surgery;
* 5. Allergic to capecitabine or oxaliplatin, or metabolic disorders;
* 6. Patients accepted Preoperative chemotherapy, radiotherapy or targeted therapy;
* 7. Attending other drug clinical trials;
* 8. Patients with Serious liver disease (such as cirrhosis, etc.), kidney disease, respiratory disease or uncontrolled diabetes, hypertension and other chronic systemic diseases, heart disease with Clinical symptoms（such as congestive heart failure, coronary heart disease symptoms, drug is difficult to control arrhythmia, hypertension, or six months had a myocardial infarction attack, or cardiac insufficiency）;
* 9. Patients with peripheral nervous system disorder or apparent mental disorders or had the history of central nervous system disorders;
* 10. Patients with serious infection(above CTCAE grade 2);
* 11. Patient with history of another malignant cancer within past 5 years（not including: cervical carcinoma in situ, non melanoma skin cancer and superficial bladder tumor );
* 12. Have the history of organ transplantation, Or have received systemic steroid therapy for a long time (note: short term user stopping medication >2 weeks can be included);
* 13. Pregnant or lactating women, women of child-bearing potential, unwilling to use adequate contraceptive protection during the process of the study;
* 14. Patients without legal capacity,or medical/ethical reasons may influence the study to continue.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2017-12-20 (Estimated); Primary Completion 2020-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival(DFS) | 5 years
  Disease Free Survivalof the Participants

SECONDARY OUTCOMES:
Overall Survival(OS) | 8 years
  Overall Survival of the Participants
Percentage of Participants With Adverse Events | 5 years
  Percentage of Participants With Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Han Liang, Master, Study Chair — Tianjin Medical University Cancer Institute and Hospital